CLINICAL TRIAL: NCT02029430
Title: An Open-Label Pilot Phase 2 Study to Investigate Efficacy, Safety, and Intratumoral Kinetics of ALDOXORUBICIN in HIV-Infected Patients With Kaposi's Sarcoma
Brief Title: A Study to Investigate ALDOXORUBICIN in HIV-infected Subjects With Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P2-KS-01
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2016-10

CONDITIONS: Kaposi's Sarcoma; HIV Positive; AIDS
Keywords: HIV positive; AIDS; Kaposi's sarcoma; Sarcoma; tumor; cancer
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Seropositivity; Acquired Immunodeficiency Syndrome; Sarcoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 mg/m2 aldoxorubicin (Experimental)
  Interventions: Drug: 50 mg/m2 aldoxorubicin
- 100 mg/m2 aldoxorubicin (Experimental)
  Interventions: Drug: 100 mg/m2 aldoxorubicin
- 150 mg/m2 aldoxorubicin (Experimental)
  Interventions: Drug: 150 mg/m2 aldoxorubicin

INTERVENTIONS:
Drug: 50 mg/m2 aldoxorubicin
  Arms: 50 mg/m2 aldoxorubicin
Drug: 100 mg/m2 aldoxorubicin
  Arms: 100 mg/m2 aldoxorubicin
Drug: 150 mg/m2 aldoxorubicin
  Arms: 150 mg/m2 aldoxorubicin

SUMMARY:
This is a pilot study to determine the efficacy, kinetics and safety of aldoxorubicin in HIV positive subjects with Kaposi's sarcoma.

DETAILED DESCRIPTION:
This is an open-label pilot phase 2 study to investigate efficacy, safety, and intratumoral kinetics of aldoxorubicin in HIV-Infected patients with Kaposi's sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age; male or female.
2. HIV (confirmed by ELISA and western blot) with histologically confirmed KS.
3. Willing to undergo serial tumor biopsies.
4. Capable of providing informed consent and complying with trial procedures.
5. KPS ≥70 (Appendix B)
6. Easter Cooperative Oncology Group (ECOG) PS 0-2.
7. Life expectancy ≥ 8 weeks.
8. Measurable (at accessible site or radiographic) tumor lesions according to ACTG TIS criteria.
9. Women must not be able to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. (Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.)
10. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
11. Geographic accessibility to the site.

Exclusion Criteria:

1. Prior exposure to an anthracycline.
2. Surgery and/or radiation treatment < 4 weeks prior to Randomization.
3. Exposure to any investigational agent within 30 days of Randomization.
4. History of other malignancies (except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix) unless documented free of cancer for ≥3 years.
5. Laboratory values: Screening serum creatinine >1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) > 2.5 × ULN, total bilirubin >1.5 × ULN, absolute neutrophil count (ANC) <1,500/mm3, platelet concentration <75,000/mm3, absolute lymphocyte count <1000/mm3, hematocrit level <25% for females or <27% for males, serum albumin ≤2.5 g/dL.
6. Evidence of central nervous system (CNS) hemorrhage National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 (published 28 May 2009) grade 2 or greater on baseline MRI.
7. Clinically evident congestive heart failure (CHF) > class II of the New York Heart Association (NYHA) guidelines.
8. Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
9. History or signs of active coronary artery disease with or without angina pectoris.
10. Serious myocardial dysfunction defined as ultrasound-determined absolute left ventricular ejection fraction (LVEF) <45% of predicted institutional normal value.
11. Active, clinically significant serious infection requiring treatment with antibacterial, antiviral (other than antiretroviral therapy), or antifungal therapy.
12. Major surgery within 4 weeks prior to Randomization.
13. Any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
14. Any condition that is unstable and could jeopardize the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Louisiana State University Health Science Center, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg/m^2 Aldoxorubicin: 50 mg/m^2 aldoxorubicin
- 100 mg/m2 Aldoxorubicin: 100 mg/m2 aldoxorubicin
- 150 mg/m^2 Aldoxorubicin: 150 mg/m^2 aldoxorubicin
Period: Overall Study
Arm/Group | 50 mg/m^2 Aldoxorubicin | 100 mg/m2 Aldoxorubicin | 150 mg/m^2 Aldoxorubicin
Started | 1 | 7 | 7
Completed (Completed defined as receiving at least one dose of study drug.) | 1 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 100 mg/m^2 Aldoxorubicin: 100 mg/m^2 aldoxorubicin
- Total: Total of all reporting groups
Arm/Group | 50 mg/m^2 Aldoxorubicin | 100 mg/m^2 Aldoxorubicin | 150 mg/m^2 Aldoxorubicin | Total
Number analyzed (Participants) | 1 | 7 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (NA) — Standard Deviation is not calculable for 1 participant | 36.7 (10.44) | 38.3 (10.87) | 38.7 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 7 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 6 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 3 | 8
  White | 1 | 2 | 4 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
HIV-Infected Patients with Kaposi's Sarcoma [Count of Participants; unit: Participants] | 1 | 7 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: To evaluate the uptake of aldoxorubicin into the tumor and the objective response rate (complete and partial response) using RECIST 1.1 criteria in subjects with HIV-infected with Kaposi's sarcoma.
  Objective responses will be evaluated using the RECIST 1.1 criteria. Changes (i.e. improvements) in tumor measurements from baseline values will be assigned a status of CR or PR or SD. Objective response measurements will comprise the sum of CR plus PR.
  Complete Response (CR): disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm).
  Partial Response (PR): 30% decrease in the sum of the longest diameter of target lesions, from the baseline sum longest diameter.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/m^2 Aldoxorubicin | 100 mg/m^2 Aldoxorubicin | 150 mg/m^2 Aldoxorubicin
Number analyzed (Participants) | 1 | 7 | 7
Participants | 0 | 7 | 6

2. Primary Outcome: Number of Participants With Treatment-related Toxicities (Adverse Events) in This Subject Population
Description: All subjects who receive any amount of ALDOXORUBICIN will be included in the safety analyses, which will include the following:
  The incidence, severity, duration, causality, seriousness, and type of AEs and changes in the subject's physical examination, vital signs, and clinical laboratory results.
  * vitals signs (systolic/diastolic blood pressure, pulse, respiration, temperature, weight, and body surface area)
  * physical examination
  * laboratory tests (chemistry, hematology, urinalysis, anion gap)
Time Frame: 30 days from last dose, up to 199 days
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg/m^2 Aldoxorubicin | 100 mg/m^2 Aldoxorubicin | 150 mg/m^2 Aldoxorubicin
Number analyzed (Participants) | 1 | 7 | 7
Participants | 1 | 6 | 6

ADVERSE EVENTS:
Time Frame: All AEs that occurred after any administration of the study medication were to be followed until the event resolved, until the subject began alternative treatment, or until the end of the study. All SAEs that occurred during the course of the study or within 30 days of the last administration, up to 199 days.
Arm/Group | 50 mg/m^2 Aldoxorubicin | 100 mg/m^2 Aldoxorubicin | 150 mg/m^2 Aldoxorubicin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/7 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/7 | 3/7
Other Adverse Events (participants affected / at risk) | 1/1 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg/m^2 Aldoxorubicin (N=1) | 100 mg/m^2 Aldoxorubicin (N=7) | 150 mg/m^2 Aldoxorubicin (N=7)
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acquired immunodeficiency syndrome (Infections and infestations) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg/m^2 Aldoxorubicin (N=1) | 100 mg/m^2 Aldoxorubicin (N=7) | 150 mg/m^2 Aldoxorubicin (N=7)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0
Medical device complication (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 3
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incision site infection (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine amniotransferase increased (Investigations) | 0 | 0 | 1
Blood HIV RNA increased (Investigations) | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0
Blood urine (Investigations) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 0
Monocyte count increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 2
Chromaturia (Renal and urinary disorders) | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT02029430/Prot_SAP_000.pdf